CLINICAL TRIAL: NCT04837963
Title: Does Hirschsprung Disease Increase the Risk of Febrile Urinary Tract Infection in Children ? A Case-control Study
Brief Title: Does Hirschsprung Disease Increase the Risk of Febrile Urinary Tract Infection in Children
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0225
Record Dates: First submitted 2021-04-06; First posted 2021-04-08 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-10

CONDITIONS: Hirschsprung Disease; Febrile Urinary Tract Infection (Disorder)
Keywords: Pediatric Surgery; Case Control study
MeSH Terms: conditions — Hirschsprung Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Febrile urinary tract infection (FUTIs) are the most common bacterial infections in children under the age of 2 years. They represent 7% of children presenting with fever without a source. In case of recurrent or undertreated FUTIs there is a risk for kidney function with the threat of chronic renal failure [7]. They are more often isolated but some FUTIs may reveal an underlying and facilitating condition. Beside the well-known congenital anomalies of the kidneys and urinary tract such as reflux or obstructions, others risk factors for FUTI are reported. Age less than 1 year, uncircumcised males, poor fluid intake, bladder bowel dysfunction (BBD) including dysfunctional voiding pattern and constipation increase the risk of FUTI. The prevalence of BBD in children with FUTIs is far higher than in the general population. Recommendations emphasize on an efficient treatment of BBD in the first-line management of recurring FUTIs and it has been proven to be efficient (ref).

One of the BBD may include Hirschsprung's Disease (HD). HD is the first congenital malformation of the enteric nervous system with a reported prevalence of 1 in 5000 live birth. It's characterized by an aganglionosis and subsequent dysmotility affect by always the anal canal, most commonly there is a rectosigmoid form (74-80%), and less commonly involves a long segment of colon (12-22%) or a total colonic aganglionosis with ileal involvement upto 50 cm proximal to ileocecal junction (4-13%). The treatment is based on the resection of dysfunctional segment of colon with an anastomosis between the normally innervated bowel to the anus, while preserving normal sphincter function. But significant bowel dysfunction may persist postoperatively. 20% of the children present a fecal incontinence, and 14% a constipation in long-term studies. Bladder dysfunction and associated urological anomalies are also reported in these patients. All of that may facilitate the occurrence of febrile urinary tract infections (FUTI) in patients with HD. Unfortunately, few studies focused on this specific population.

The objective of this study was to find out whether children with HD are more prone to develop FUTIs than controls and which patient with HD are more at risk to develop UTIs.

ELIGIBILITY:
Inclusion criteria:

Patients :

- surgical treatment of an HD confirmed on histopathologic exam.

Controls :

- appendicetomy for acute appendicitis without history of HD, ano rectal malformation or any other colic disease

Exclusion criteria:

* patients with HD but not yet operated
* patient with a stoma at the time of the study
* patient with chronic intestinal pseudo obstruction without HD

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Cases were patients who underwent surgical treatment of an HD confirmed on histopathologic exam. Controls were children who underwent an appendicetomy for acute appendicitis without history of HD, ano rectal malformation or any other colic disease.. Two controls were matched for age and sex, at least included for each case
Sampling Method: Non-Probability Sample
Enrollment: 630 (Actual)
Dates: Start 2021-05-16 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
Compare the risk of febril urinary tract infection | Day 1
  Compare the risk of febril urinary tract infection between children with Hirschsprung disease and control Febrile urinary tract infection was defined as a positive urine examination with a single bacteria with more than 10.5 cfu/mL and more than 10.4 leukocytes/ml associated with fever above 38.5°C and C-reactive protein (CRP) above 50 mg/

SECONDARY OUTCOMES:
Compare the age at the time of febrile urinary tract infection | Day 1
  Compare the age at the time of febrile urinary tract infection between children with Hirschsprung disease and control. This event could occur sooner in children with Hirschsprung disease than controls.
Febrile urinary tract infection risk factor | Day 1
  Febrile urinary tract infection risk factor for children with Hirschsprung disease based upon the form of the disease, kinf of surgery, functional results For each patient treated by Hirschsprung disease, surgical technique, the level of involvement and the functional outcome will be collected.
  The functional outcome was evaluated through the number of stool per day, the presence of soiling, the need of additional antegrade or retrograde colonic enema

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas KALFA, Study Director — University Hospital, Montpellier
Locations (1):
- University hospital of Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC